CLINICAL TRIAL: NCT05115071
Title: The Effect of Online Childbirth Preparation Education in Pregnancy on Worries and Fear of Birth, Preparation for Birth, and Well-being of Self and Baby in the Covid 19 Pandemic
Brief Title: Online Childbirth Preparation Education in Covid-19 Pandemic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Okan Vardar, Lecturer, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-60116787-020-10516
Record Dates: First submitted 2021-11-06; First posted 2021-11-10 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Birth, First; COVID-19; Fear of Childbirth
Keywords: online childbirth preparation; fear of childbirth; worries on birth; preparation for birth; well-being of self and baby; Covid 19 pandemic
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Single blind pre-post test randomized controlled design
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental)
  Interventions: Behavioral: Childbirth preparation education
- No intervention (No Intervention)

INTERVENTIONS:
Behavioral: Childbirth preparation education — Purpose: The aim of the birth preparation education is to eliminate the fears and concerns of pregnant women about birth and to prepare them for birth during the Covid-19 Pandemic process.
  Education hours: The education will be completed in total two weeks and eight hours, consisting of two days and four hours each week.
  Method: The education will be given online through the Microsoft Teams application. Each training day will consist of two lessons. Each lesson will last 45 minutes. There will be a 15-minute break between the two lessons. The first lesson will be conducted in the form of a question and answer session with a power-point presentation.In the second lesson, relaxation exercises will be applicated and evaluations will be taken at the end of the lesson.
  The group that will receive the education: Healthy pregnant women between 24-34 weeks of gestation will be included in the training. Trainings will continue with closed groups.
  Arms: Experimental

SUMMARY:
Today, pregnancy and childbirth are important life events that involve many difficulties and changes that must be overcome for both men and women. During this process, changes occur in the pregnant woman's body, emotional state and family life. These changes often cause pregnant women to experience anxiety about the baby's health and their own health, and to create new stressful situations. Adding the pandemic conditions to this situation further complicates the process and it is seen that the fears of women towards the birth and postpartum period will increase even more. Childbirth preparation classes reduce the fear and anxiety of women and create a positive perception of birth. For this reason, it is more important to give birth preparation education to women during in pregnancy during the pandemic period. However, it is not possible to give face-to-face birth preparation education to women in this process. For this reason, the aim of this study is to examine the effect of online childbirth preparation education in pregnancy on worries and fear of birth, preparation for birth, and well-being of self and baby in the Covid 19 pandemic.

The research is a pre-post test randomized controlled experimental study. The block randomization method will be used. The universe of the research will consist of women who applied to Pamukkale University Research and Application Hospital pregnant outpatient clinic, and have a healthy pregnancy at 24-34 weeks of gestation. The education will be done online. The sample size was calculated in the G*power statistics program using the data of a study in which the childbirth preparation education intervention was previously performed (α =0.05, d=1.05). Accordingly, it was found that 16 people should be taken for each group to sampling for 80% power. Considering that there might be losses, the number of samples was increased by 10% and it was planned to include a total of 36 people in the study. Intention-to-treat analysis will be performed to manage bias and losses.

ELIGIBILITY:
Inclusion Criteria:

* Be over 18 years old
* Volunteering to participate in research
* Be at 24-34 weeks of gestation
* Be nulliparous
* Not having a high risk pregnancy
* Be able to read and write Turkish
* Be able to fill out an online survey form
* Planning to have a normal spontaneous vaginal delivery

Exclusion Criteria:

* Be under the age of 18
* Not completing eight hours of childbirth preparation education
* Having a mental disorder that prevents answering survey questions
* Having a psychiatric illness
* Be able not use Microsoft Teams app

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant women
Enrollment: 44 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2021-11-25 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Oxford Worries on Labour Scale (OWLS) | Change from baseline Oxford Worries on Labour score at 2 weeks
  The scale will be filled online by each pregnant woman before and after the education. The scale is used to evaluate concerns about the birth process and consists of 10 items. Scoring is done between 1-4. The scale consists of 3 sub-dimensions. There is no reverse scored item. The points that can be taken are min:10, max:40. As the score increases, it is interpreted that the anxiety level of women decreases.
Prenatal Self Evaluation Questionnaire (PSEQ)-Preparation for labor subscale | Change from baseline Preparation for Labor score at 2 weeks
  The scale will be filled online by each pregnant woman before and after the education. The scale was developed to evaluate the adaptation of women in the prenatal period to motherhood. The scale consists of 7 sub-dimensions and a total of 79 items. Scoring is done between 1-4. Items 7, 13, 24, 25, 26, 38, 47, 48, 56, 72 belong to the Preparation for Labor subscale. There are reversed items in the scale. Low scores indicate high compliance to pregnancy.
Prenatal Self Evaluation Questionnaire (PSEQ)-Well-being of self and baby subscale | Change from baseline Well-being of Self and Baby score at 2 weeks
  The scale will be filled online by each pregnant woman before and after the education.The scale was developed to evaluate the adaptation of women in the prenatal period to motherhood. The scale consists of 7 sub-dimensions and a total of 79 items. Scoring is done between 1-4. The scale was developed to evaluate the adaptation of women in the prenatal period to motherhood. The scale consists of 7 sub-dimensions and a total of 79 items. Scoring is done between 1-4. Items 12, 16, 17, 30, 41, 51, 57, 63, 68, 71 belong to the Well-Being of Self and Baby subscale. There are reversed items in the scale. Low scores indicate high compliance with pregnancy.
Fear of Birth Scale (FOBS) | Change from baseline Fear of Birth score at 2 weeks
  The scale will be filled online by each pregnant woman before and after the education. The scale was developed to measure the fear of childbirth. In the scale, the participants asked the question "How do you feel about the upcoming birth right now?" In response to the question, they are asked to rate their emotions by marking them on two 100 mm lines defined as (a) 'calm and anxious', (b) 'no fear and severe fear'. The cut-off point of the scale is 50 points. It has been defined that people who score 50 and above experience fear of childbirth. The scale can be applied to both pregnant women and their partners. Scoring of the scale: The scores marked on two 100 mm lines are summed and divided into two. The resulting score gives the FOBS score of the pregnant or spouse who answered the scale. Individuals with a score of 50 and above are considered to have fear of childbirth.
The Fear of COVID-19 Scale (FCV-19S) | Change from baseline Fear of Covid-19 score at 2 weeks
  The scale will be filled online by each pregnant woman before and after the education. The scale is used to measure fear of Covid-19. The scale consists of one dimension and 7 items. Scoring is done between 1-5. There is no reverse scored item. The points that can be taken are min:7, max:35. An increase in the score obtained from the scale means an increase in the fear of Covid-19.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)